CLINICAL TRIAL: NCT00798070
Title: A Randomised Phase 3 Study Comparing Biweekly and Tailored Epirubicin + Cyclophosphamide Followed by Biweekly Tailored Docetaxel Versus Three Weekly Epirubicin + Cyclophosphamide + 5-fluorouracil Followed by Docetaxel in Lymph Node Positive or High Risk Lymph Node Negative Breast Cancer Patients
Brief Title: Panther: A Study Comparing Biweekly and Tailored EC-T Versus Three Weekly FEC-T in Breast Cancer Patients
Acronym: PANTHER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Swedish Breast Cancer Group (Other); Austrian Breast & Colorectal Cancer Study Group (Network); GBG Forschungs GmbH (Other)
Responsible Party: Principal Investigator, Prof Jonas Bergh, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANTHER SBG2004-1; 2007-002061-12 (EudraCT Number); ISRCTN39017665 (Registry Identifier: ISRCTN); ABCSG25 (Other: Austrian Breast and Colorectal Cancer Study Group); GBG53 (Other: German Breast Group)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Lymph node positive or high risk lymph node negative breast; cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: dtEC→dtT (Experimental): Individually tailored and two weekly dosed epirubicin + cyclophosphamide followed by a three weeks break followed by biweekly and tailored docetaxel (dtEC→dtT) given every second week
  Interventions: Drug: dtEC→dtT
- Arm B: FEC→T (Active Comparator): Fixed dosed and three weekly epirubicin, cyclophosphamide and 5-fluorouracil, followed by fixed dosed and three weekly docetaxel
  Interventions: Drug: FEC→T

INTERVENTIONS:
Drug: dtEC→dtT — Individually tailored and two weekly dosed epirubicin (start dose 90mg/m2) + cyclophosphamide (start dose 600mg/m2) followed by a three weeks break followed by biweekly and tailored docetaxel (start dose 75mg/m2) given every second week. If toxicity measured by CTC-NCI criteria are grade 2 or less (except haematological toxicity) it will be possible to escalate doses
  Other Names: Epirubicin; Cyclophosphamide; Taxotere
  Arms: Arm A: dtEC→dtT
Drug: FEC→T — Fixed dosed and three weekly epirubicin (100mg/m2), cyclophosphamide (500mg/m2) and 5-fluorouracil (500mg/m2), followed by fixed dosed and three weekly docetaxel (100mg/m2), no dose escalations.
  Other Names: Epirubicin; Cyclophosphamide; Fluorouracil; Taxotere
  Arms: Arm B: FEC→T

SUMMARY:
This is an adjuvant, open, prospective, randomized study to compare:

A. Individually tailored and two weekly dosed epirubicin + cyclophosphamide followed by a three weeks break followed by biweekly and tailored docetaxel (dtEC→dtT) given every second week, to

B. Fixed dosed and three weekly epirubicin, cyclophosphamide and 5-fluorouracil, followed by fixed dosed and three weekly docetaxel (FEC→T).

Patients with primary node-positive or high risk lymph node negative breast cancer will be eligible for the study.

The primary objective of the phase 3 study is to compare breast cancer relapse-free survival (BCRFS) between the dtEC→dtT and FE100C→T. To detect a five-year BCRFS difference of 0.710 to 0.790 about 1000 patients per arm will be needed. They will be recruited during four years and followed another two years for breast cancer events.

Secondary objectives are to compare

1. Distant disease-free survival (DDFS)
2. Event-free survival and
3. Overall survival
4. Health-related quality of life and toxicity analyses according to CTC
5. Outcome in relation to tumour biological factors and polymorphism patterns

   1. RFS in relation to the Sorlie classes using immunohistochemical markers and/or gene expression profiling comparing A vs B arm
   2. RFS with receptor positive disease (analyzed in the local laboratories as described in the CRFs and also analyzed as continuous variables) in the comparison between the A- and B- arms.
   3. RFS with high and low proliferation, respectively, (analyzed in the local laboratories as described in the CRFs and also analyzed as a continuous variable, or centrally analyzed), in the comparison between the A- and B-arms.
   4. RFS in relation to HER-2/neu status (analyzed in the local laboratories as described in the CRFs) in the primary cancers in the comparison between the A- and B-arms and analyzed whether trastuzumab was given in sequence or concurrently.
   5. RFS analyzed in relation to other molecular markers (e.g. gene expression profiling/ sequencing) in the primary cancers and SNPs signatures in normal DNA (related to toxicities for EC/FEC and docetaxel components, respectively, and given dose levels and outcome in relation to these factors and in relation QoL) to outcome per arm.
   6. RFS analyzed in relation to tumour associated lymphocytes and Y-box binding protein in the comparison between the A- and B-arms.

Tumour tissue will be obtained and stored for studies of prognostication and therapy prediction.

Last patient randomized was September 2011.

DETAILED DESCRIPTION:
Are described under the heading "Outcome measures"

ELIGIBILITY:
Inclusion Criteria:

* Histological proven invasive primary breast cancer, with at least 5 (recommended 10) removed axillary lymph nodes OR negative sentinel node biopsy performed for the node negative cohort. Interval between definitive surgery that includes axillary lymph node dissection and registration must be less than 60 days. Paraffin block from the primary tumour must be retained (not mandatory for Austrian sites). Frozen tumour tissue is strongly recommended to be stored.
* Receptor negative or positive tumours with 1 or more positive axillary lymph nodes (more than 0.2 mm) OR axillary node negative breast cancers if the primary tumour is larger than 20 mm and receptor negative (Er and Pgr with no receptor content) and being Elston grade III. In Germany high risk node negative breast cancer patients are not eligible until labelling for docetaxel includes node-negative disease.
* A primary breast cancer patient being 35 years or younger considered suitable for adjuvant chemotherapy (may be receptor negative or positive, HER-2/neu negative or positive, with or without axillary lymph node metastases).
* Macroscopically and microscopically free margins after radical surgery (no cancer cells at borders of resection).
* No proven distant metastases (negative chest/pulmonary X-ray, bone scintigram (when clinical signs of skeletal metastases or elevated ALP) supplemented with normal conventional X-ray of hot spots, normal liver function test and haematological function tests; when abnormal values, CT or ultrasound of the liver, patient can be included if no metastases are demonstrated.
* Female age 18-65.
* Ambulant patients (ECOG 1 or less).
* No major cardiovascular morbidity NYHA I or II. (Appendix 3).
* Written informed consent according to the local ethics committee requirements.
* Patients of childbearing potential should have a negative pregnancy test within seven days of registration. (In Austria, pregnancy tests have to be repeated monthly during the treatment phase).

Exclusion Criteria:

* Previous neo-adjuvant treatment.
* Non-radical surgery (histopathological positive margins).
* Proven distant metastases.
* Pregnancy or lactation.
* Other serious medical condition.
* Previous or concurrent malignancies at other sites, except basal cell carcinoma and/or squamous cell carcinoma in situ of the skin or cervix. Patients with previous breast cancer (invasive and/or ductal carcinoma in situ) in the other breast without loco-regional (large lung volumes) radiotherapy, without objective findings for relapse, with > 5 years since diagnosis can be included.
* Abnormal laboratory values precluding the possibility to safely deliver the used cytotoxic agents in the study.
* Hypersensitivity to drugs formulated in polysorbate 80.
* Peripheral neuropathy grade ≥2.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2017 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Breast cancer relapse-free survival | 2 years
  Breast cancer recurrence free survival is defined as time from randomization to the first of the events; local-, regional- or distant breast cancer recurrence or death due to breast cancer or last date of follow-up if no event has occurred. This was defined already in the phase 2 protocol (1 Sept 2004).

SECONDARY OUTCOMES:
Distant disease-free survival | 2 years
  Distant disease free survival is defined as time from randomization to the first of distant metastases or death due to breast cancer.
Event-free survival | 2 years
  Event-free survival is defined as time from randomization to the first of the events breast cancer recurrence (any type), contra-lateral breast cancer, other malignancy or any cause of death.
Overall survival | 2 years
  Overall survival is defined as time from randomization to any death.
Health-related quality of life and toxicity analyses according to CTC | 2 years
Outcome in relation to tumour biological factors and polymorphism patterns | 2 years
  Comparing arm A vs B regarding:
  1. RFS in relation to the Sorlie classes using immunohistochemical markers and/or gene expression profiling comparing A vs B arm;
  2. RFS with receptor positive disease in the comparison between the A- and B arms;
  3. RFS with high and low proliferation, respectively, in the comparison between the A- and B-arms.;
  4. RFS in relation to HER-2/neu status in the primary cancers in the comparison between the A- and B-arms and analyzed whether trastuzumab was given in sequence or concurrently;
  5. RFS analyzed in relation to other molecular markers in the primary cancers and SNPs signatures in normal DNA to outcome per arm;
  6. RFS analyzed in relation to tumour associated lymphocytes and Y-box binding protein in the comparison between the A- and B-arms.
  Description of a to e are more detailed in the protocol, shortened here due to space limitation.
BCRFS in arm A in relation to given dose levels | 2 years
  Breast cancer relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Bergh, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (80):
- Austria (10):
  - MUG - Med. Univ.-Klinik Graz, Graz
  - MUI - Univ. Klinik f. Frauenheilkunde, Innsbruck, Innsbruck
  - LKH Leoben, Leoben
  - AKH Linz, Linz
  - KH BHS Linz, Linz
  - LKH Rankweil, Rankweil
  - KH BHB St. Veit/Glan, Saint Veit/Glan
  - LKH Salzburg / PMU, Salzburg
  - Brustzentrum Hanusch-KH, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Germany (59):
  - Marienhospital, Aachen
  - Klinikum am Bruderwald, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - HELIOS Klinikum, Berlin
  - Klinikum Bietigheim, Bietigheim
  - Johanniter Krankenhaus, Bonn
  - Universitätsfrauenklinik, Bonn
  - Klinikum Sindelfingen-Böblingen, Böblingen
  - Krankenhaus Celle, Celle
  - St. Elisabeth-KKH, Cologne
  - Klinikum Deggendorf, Deggendorf
  - Diakonissen Krankenhaus, Dresden
  - Gemeinschaftspraxis, Dresden
  - Krankenhaus St. Joseph-Stift, Dresden
  - Praxis Dr. Adhami, Erkelenz
  - Klinikum der J. W. Goethe Universität, Frankfurt am Main
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Onkologische Gemeinschaftspraxis, Frankfurt am Main
  - Kreiskrankenhaus, Freudenstadt
  - Klinikum Fulda, Fulda
  - Onkologische Schwerpunktpraxis, Goslar
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - Universitätsfrauenklinik, Halle
  - Klinikum Hameln, Hamelin
  - Henriettenstiftung, Hanover
  - Medizinische Hochschule, Hanover
  - Universität Heidelberg, Heidelberg
  - Klinikum Heilbronn, Heilbronn
  - Gemienschaftspraxis, Hildesheim
  - Universitätsfrauenklinik, Homburg
  - St. Vincentius Kliniken, Karlsruhe
  - Städtisches Klinikum, Karlsruhe
  - Elisabeth Krankenhaus, Kassel
  - Klinikum Kempten, Kempten
  - St. Vincenz Krankenhaus, Limburg
  - Onkologische Tagesklinik, Lohsa
  - Klinikum Ludwigsburg, Ludwigsburg
  - Ev. Krankenhaus, Ludwigsfelde
  - St. Vincenz und Elisabeth-Hospital, Mainz
  - Universitätsfrauenklinik, Mainz
  - Universitätsfrauenklinik, Mannheim
  - Klinikum Fichtelgebirge, Marktredwitz
  - Onkologische Praxis, Memmingen
  - Gemeinschaftspraxis Münster, Münster
  - Praxis am Klinikum Neumarkt, Neumarkt
  - Onkologische Praxis, Pinneberg
  - Klinikum am Steinenberg, Reutlingen
  - Klinikum Rheinfelden, Rheinfelden
  - Klinikum Schwerin, Schwerin
  - Gesellschaft für onkologische Studien, Troisdorf
  - Klinikum Tuttlingen, Tuttlingen
  - Universitätsfrauenklinik, Tübingen
  - Universitätsfrauenklinik, Ulm
  - Klinikum Villingen-Schwenningen, Villingen
  - Klinikum Weiden, Weiden
  - Klinikum Weinheim, Weinheim
  - Asklepios Paulinen Klinik, Wiesbaden
  - St. Josefs-Hospital, Wiesbaden
  - Stadtkrankenhaus, Worms
- Sweden (11):
  - Central Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Central Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Malmö General University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Dept of Oncology, Stockholm
  - Central Hospital, Sundsvall
  - Norrlands University Hospital, Umeå
  - Uppsala Academic Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Oral presentation at ASCO 4 June 2016 (completed).

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Increasing the dose intensity of chemotherapy by more frequent administration or sequential scheduling: a patient-level meta-analysis of 37 298 women with early breast cancer in 26 randomised trials. Lancet. 2019 Apr 6;393(10179):1440-1452. doi: 10.1016/S0140-6736(18)33137-4. Epub 2019 Feb 8. PMID 30739743
- [Result] Matikas A, Papakonstantinou A, Loibl S, Steger GG, Untch M, Johansson H, Tsiknakis N, Hellstrom M, Greil R, Mobus V, Gnant M, Bergh J, Foukakis T. Benefit from dose-dense adjuvant chemotherapy for breast cancer: subgroup analyses from the randomised phase 3 PANTHER trial. Lancet Reg Health Eur. 2024 Dec 3;49:101162. doi: 10.1016/j.lanepe.2024.101162. eCollection 2025 Feb. PMID 39703564
- [Result] Matikas A, Mobus V, Greil R, Andersson A, Steger GG, Untch M, Fornander T, Malmstrom P, Schmatloch S, Johansson H, Hellstrom M, Brandberg Y, Gnant M, Loibl S, Foukakis T, Bergh J; SweBCG, ABCSG and GBG. Tailored Dose-Dense Versus Standard Adjuvant Chemotherapy for High-Risk Early Breast Cancer: End-of-Study Results of the Randomized PANTHER Trial. J Clin Oncol. 2024 Sep 10;42(26):3077-3082. doi: 10.1200/JCO.24.00178. Epub 2024 Jul 17. PMID 39018515
- [Result] Zerdes I, Simonetti M, Matikas A, Harbers L, Acs B, Boyaci C, Zhang N, Salgkamis D, Agartz S, Moreno-Ruiz P, Bai Y, Rimm DL, Hartman J, Mezheyeuski A, Bergh J, Crosetto N, Foukakis T. Interplay between copy number alterations and immune profiles in the early breast cancer Scandinavian Breast Group 2004-1 randomized phase II trial: results from a feasibility study. NPJ Breast Cancer. 2021 Nov 19;7(1):144. doi: 10.1038/s41523-021-00352-3. PMID 34799582
- [Result] Brandberg Y, Johansson H, Hellstrom M, Gnant M, Mobus V, Greil R, Foukakis T, Bergh J; Swedish Breast Cancer Group, the Austrian Breast, Colorectal Cancer Study Group, the German Breast Cancer Group. Long-term (up to 16 months) health-related quality of life after adjuvant tailored dose-dense chemotherapy vs. standard three-weekly chemotherapy in women with high-risk early breast cancer. Breast Cancer Res Treat. 2020 May;181(1):87-96. doi: 10.1007/s10549-020-05602-9. Epub 2020 Mar 31. PMID 32232698
- [Result] Papakonstantinou A, Matikas A, Bengtsson NO, Malmstrom P, Hedayati E, Steger G, Untch M, Hubbert L, Johansson H, Hellstrom M, Gnant M, Loibl S, Greil R, Moebus V, Foukakis T, Bergh J. Efficacy and safety of tailored and dose-dense adjuvant chemotherapy and trastuzumab for resected HER2-positive breast cancer: Results from the phase 3 PANTHER trial. Cancer. 2020 Mar 15;126(6):1175-1182. doi: 10.1002/cncr.32653. Epub 2019 Dec 18. PMID 31851385
- [Result] Papakonstantinou A, Hedayati E, Hellstrom M, Johansson H, Gnant M, Steger G, Greil R, Untch M, Moebus V, Loibl S, Foukakis T, Bergh J, Matikas A. Neutropenic complications in the PANTHER phase III study of adjuvant tailored dose-dense chemotherapy in early breast cancer. Acta Oncol. 2020 Jan;59(1):75-81. doi: 10.1080/0284186X.2019.1670353. Epub 2019 Oct 4. PMID 31583943
- [Result] Matikas A, Foukakis T, Moebus V, Greil R, Bengtsson NO, Steger GG, Untch M, Johansson H, Hellstrom M, Malmstrom P, Gnant M, Loibl S, Bergh J. Dose tailoring of adjuvant chemotherapy for breast cancer based on hematologic toxicities: further results from the prospective PANTHER study with focus on obese patients. Ann Oncol. 2019 Jan 1;30(1):109-114. doi: 10.1093/annonc/mdy475. PMID 30357310
- [Result] Matikas A, Margolin S, Hellstrom M, Johansson H, Bengtsson NO, Karlsson L, Edlund P, Karlsson P, Lidbrink E, Linderholm B, Lindman H, Malmstrom P, Villman K, Foukakis T, Bergh J. Long-term safety and survival outcomes from the Scandinavian Breast Group 2004-1 randomized phase II trial of tailored dose-dense adjuvant chemotherapy for early breast cancer. Breast Cancer Res Treat. 2018 Apr;168(2):349-355. doi: 10.1007/s10549-017-4599-4. Epub 2017 Nov 30. PMID 29190004
- [Result] Foukakis T, von Minckwitz G, Bengtsson NO, Brandberg Y, Wallberg B, Fornander T, Mlineritsch B, Schmatloch S, Singer CF, Steger G, Egle D, Karlsson E, Carlsson L, Loibl S, Untch M, Hellstrom M, Johansson H, Anderson H, Malmstrom P, Gnant M, Greil R, Mobus V, Bergh J; Swedish Breast Cancer Group (SweBCG), the German Breast Group (GBG), and the Austrian Breast & Colorectal Cancer Study Group (ABCSG). Effect of Tailored Dose-Dense Chemotherapy vs Standard 3-Weekly Adjuvant Chemotherapy on Recurrence-Free Survival Among Women With High-Risk Early Breast Cancer: A Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1888-1896. doi: 10.1001/jama.2016.15865. PMID 27825007
- [Result] Bergh J. Oral presentation, ASCO Annual Meeting 2016.
- [Result] Margolin S, Bengtsson NO, Carlsson L, Edlund P, Hellstrom M, Karlsson P, Lidbrink E, Linderholm B, Lindman H, Malmstrom P, Pettersson Skold D, Soderberg M, Villman K, Bergh J; Scandinavian Breast Group Study SBG 2004-1. A randomised feasibility/phase II study (SBG 2004-1) with dose-dense/tailored epirubicin, cyclophoshamide (EC) followed by docetaxel (T) or fixed dosed dose-dense EC/T versus T, doxorubicin and C (TAC) in node-positive breast cancer. Acta Oncol. 2011 Jan;50(1):35-41. doi: 10.3109/0284186X.2010.535847. PMID 21174610